CLINICAL TRIAL: NCT03043794
Title: A Phase II Study of Preoperative Single Fraction Stereotactic Body Radiotherapy to the Intact Breast in Early Stage Low Risk Breast Cancer: Analysis of Radiation Response
Brief Title: Study of Stereotactic Radiotherapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI closed. Unable to enroll enough patients to collect and analyze data.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Robert L. Sloan Fund for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1741; IRB00128074 (Other: JHM IRB)
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: early stage; low risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: SBRT to the breast follow by standard of care surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SBRT to the breast then surgery (Experimental): Stereotactic Body Radiation Therapy (SBRT) of 21Gy followed by standard of care surgery
  Interventions: Radiation: Stereotactic Body Radiation Therapy SBRT

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy SBRT — Stereotactic Body Radiation Therapy to the breast to 21 Gy

SUMMARY:
This is a Phase II trial of preoperative stereotactic radiation to the breast for low risk breast cancer.

DETAILED DESCRIPTION:
This is a single arm phase II study design, evaluating the pathologic response (primary endpoint) as well as toxicity, cosmetic outcome, quality of life, and translational correlates (secondary endpoints) to pre-operative stereotactic body radiotherapy (SBRT) to intact breast tumors in patients with hormone-receptor positive early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age > or = to 50 years of age
* Invasive ductal carcinoma
* Clinically and radiographically T1 tumor
* Clinically node negative
* Clearly demarcated tumor on magnetic resonance imaging (MRI), as determined by treating physician (MRI may be done after enrollment if not done prior)
* Planning breast conserving surgery including sentinel node biopsy
* ≥10% expression of ER and/or PR
* HER2- using the current College of American Pathologists guidelines
* Post-menopausal
* Willing and able to provide informed consent

Exclusion Criteria:

* Medical conditions that may increase risk for poor cosmetic outcome (i.e. Lupus, rheumatoid arthritis, scleroderma
* Pure DCIS without invasive cancer
* Patients who have received or will be receiving neoadjuvant systemic therapy, endocrine therapy, or targeted agents
* Breast implant in the involved breast unless the implant will be removed prior to initiation of study treatment
* Positive pregnancy test
* Subjects without placement of a biopsy clip at the diagnostic procedure who are unwilling to undergo clip placement.
* Unable to meet dosimetric constraints due to tumor location and/or patient anatomy
* Planning mastectomy
* Unable to tolerate prone positioning

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females only
Enrollment: 4 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2023-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wright, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT to the Breast Then Surgery: Stereotactic Body Radiation Therapy of 21Gy to the breast followed by standard of care surgery
Period: Overall Study
Arm/Group | SBRT to the Breast Then Surgery
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Stereotactic Body Radiation Therapy to the Breast Then Surgery: Stereotactic Body Radiation Therapy (SBRT) of 21 Gy to the breast, followed by standard of care surgery.
Arm/Group | Stereotactic Body Radiation Therapy to the Breast Then Surgery
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: Years] | 68.25 [60 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response Measured by Residual Cancer Burden (RCB)
Description: Number of participants with Residual Cancer Burden (RCB) designation 0 (also known as pathologic complete response (pCR)), and RCB I designation (combined endpoint of either of those designations) 4-6 weeks after pre-operative SBRT to intact breast tumors.
Time Frame: 4-6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- SBRT to the Breast Then Surgery: Stereotactic Body Radiation Therapy of 21Gy followed by standard of care surgery
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
Participants
  RCB designation 0 | 1
  RCB designation 1 | 3

2. Secondary Outcome: Number of Participants With Treatment-related Toxicity
Description: The number of participants with severe acute toxicity, defined as any CTCAE v4 grade 3 or higher toxicity noted from RT delivery up to 90 days after completion of surgery, up to 4 months.
Time Frame: RT delivery up to 90 days after completion of surgery, up to 4 months
Measure: Count of Participants; unit: Participants
Groups:
- SBRT to the Breast Then Surgery: Stereotactic Body Radiation of 21 gy followed by standard of care surgery
  Stereotactic Body Radiation SBRT: Stereotactic Body Radiation to the breast to 21 Gy
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Cosmetic Outcome (Patients)
Description: Number of patients who report poor cosmetic outcomes from patient perspective at 90 days after pre-operative SBRT to intact breast tumors using the Radiation therapy oncology group (RTOG) cosmesis scale and digital images.
  RTOG Cosmesis Scale: 1 (excellent), 2 (good), 3 (fair), and 4 (poor)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Local Recurrence
Description: To measure local recurrence in participants
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Breast Cancer Treatment Outcomes Scale (BCTOS)
Description: To assess patient reported satisfaction and quality of life with treatment using the Breast Cancer Treatment Outcomes Scale (BCTOS). The BCTOS is a questionnaire that evaluates the aesthetic and functional outcomes of breast conserving surgery (BCS). Patients rate each item on the questionnaire using a four-point Likert scale, with 1 indicating no difference and 4 indicating a large difference between the treated and untreated breast. Score range 22-88. Higher scores indicate higher difference.
Time Frame: Pre and Post surgery (Up to 3 years)
Population: Patients with data collected are reported.
Measure: Number; unit: score on a scale
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
score on a scale
  Participant 1, Pre-treamtment: number analyzed (Participants) | 1
  Participant 1, Pre-treamtment | 22
  Participant 1, Post surgery: number analyzed (Participants) | 1
  Participant 1, Post surgery | 31
  Participant 2, Pre-treatment: number analyzed (Participants) | 1
  Participant 2, Pre-treatment | 22
  Participant 2, Post surgery: number analyzed (Participants) | 1
  Participant 2, Post surgery | 23
  Participant 3, Pre-treatment: number analyzed (Participants) | 1
  Participant 3, Pre-treatment | 22
  Participant 4, Pre-treatment: number analyzed (Participants) | 1
  Participant 4, Pre-treatment | 22

6. Secondary Outcome: Cosmetic Outcome (Provider)
Description: Number of providers who report poor cosmetic outcomes from provider perspective at 90 days after pre-operative SBRT to intact breast tumors using the RTOG (Radiation therapy oncology group) cosmesis scale and digital images.
  RTOG Cosmesis Scale: 1 (excellent), 2 (good), 3 (fair), and 4 (poor)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT to the Breast Then Surgery
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | SBRT to the Breast Then Surgery
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT to the Breast Then Surgery (N=4)
Fatigue (General disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Induration (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early, only 4 participants were enrolled. Enrollment was too challenging to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03043794/Prot_SAP_000.pdf